CLINICAL TRIAL: NCT04509271
Title: Shanghai Mental Health Center
Brief Title: Study on Novel Peripheral Blood Diagnostic Biomarkers for MCI Due to Alzheimer's Disease
Acronym: Precision1000
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: WT20200808
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood plasma and non-coding RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Normal aged
  Interventions: Diagnostic Test: MicRNAs battery kits
- MCI due to AD
  Interventions: Diagnostic Test: MicRNAs battery kits
- Mild AD
  Interventions: Diagnostic Test: MicRNAs battery kits
- Moderate AD
  Interventions: Diagnostic Test: MicRNAs battery kits
- Severe AD
  Interventions: Diagnostic Test: MicRNAs battery kits
- Dementia with Lewy body
  Interventions: Diagnostic Test: MicRNAs battery kits
- Frontotemporal dementia
  Interventions: Diagnostic Test: MicRNAs battery kits

INTERVENTIONS:
Diagnostic Test: MicRNAs battery kits — Novel peripheral blood diagnostic biomarker for MCI due to AD.

SUMMARY:
The prevalence of Mild Cognitive Impairment (MCI) is about 15%-17%. 10%-15% of MCI progresses to Alzheimer's disease (AD) every year. The annual incidence of MCI in the normal elderly is about 1%. Peripheral Blood biomarkers is the key and difficult points in AD research. Except expensive brain β amyloid plaque imaging, few breakthroughs of early diagnosis technology of MCI due to AD can be made to facilitate clinical application. Even Tau-181 and Tau-217 were reported in this year on Lancet neurology and JAMA. We also need to study on the biomarkers upstream of pathological changes about senile plaque. The purpose of this program is to study the reliability and validity of plasma miRNAs for early diagnosis of MCI due to AD and other dementia such as DLB and FTLD. The clinical diagnosis of AD and MCI due to AD are according to the National Institute of Aging and the Alzheimer's Disease Association (NIA-AA) diagnostic criteria in 2011. Plaque imaging is used to be golden criteria for the diagnosis of AD and MCI due to AD.

ELIGIBILITY:
Inclusion Criteria:

* 2011 NIA-AA criteria of MCI due to AD or AD or - 2017 Diagnosis and management of dementia with Lewy bodies: Fourth consensus report of the DLB Consortium or - 2001 the McKhann consensus clinical criteria for FTD (McKhann et al.)

Exclusion Criteria:

* Dementia caused by infection or substance
* Thyroid disease

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NC, AD, DLB, FTD and MCI due to AD
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of biomarkers for MCI due to AD and other dementia. | 1 and half years
  MicRNAs battery for diagnostic of MCI due to AD

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
According to the approval of IRB.

REFERENCES:
- [Derived] Ma YM, Zhao L. Mechanism and Therapeutic Prospect of miRNAs in Neurodegenerative Diseases. Behav Neurol. 2023 Nov 23;2023:8537296. doi: 10.1155/2023/8537296. eCollection 2023. PMID 38058356